CLINICAL TRIAL: NCT02631005
Title: Walk With Ease Program For Patients With Systemic Lupus Erythematosus
Acronym: Walk SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-2738
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; exercise
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walk With Ease Participants (Experimental): Participants will receive a copy of the "Walk With Ease" workbook. This workbook provides guidance on walking safety and on how to start and maintain a regular walking program. It is designed to help participants increase their physical activity over a six-week period. Participants will complete self-reported outcomes questionnaires before and after completion of the program.
  Interventions: Other: "Walk With Ease"

INTERVENTIONS:
Other: "Walk With Ease" — Six-week walking program

SUMMARY:
The purpose of this study is to evaluate the effects of "Walk With Ease", a moderate-intensity exercise program, on pain, stiffness, and fatigue caused by lupus. Participants will receive a copy of the "Walk With Ease" workbook. The book provides guidance about walking safety as well as how to start, build-up, and maintain a walking program. Participants will complete questionnaires assessing their symptoms before and after completing the six-week program.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of "Walk With Ease", a moderate-intensity exercise program, on pain, stiffness, and fatigue caused by lupus. Participants will receive a copy of the "Walk With Ease" workbook, a publication of the Arthritis Foundation. Participants will complete self-reported outcomes questionnaires prior to beginning the program and six weeks later at completion of the program. The questionnaires will include visual analog scales for pain, stiffness, and fatigue as well as a FACIT-Fatigue form. Participants will also complete a satisfaction survey at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of systemic lupus erythematosus
* Age >/= 18

Exclusion Criteria:

* Age <18
* Engagement in >150 minutes of moderate-intensity activity at baseline
* Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score >8
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score from Baseline to Six Weeks | 6 weeks
  Pain scale ranges from 0 millimeters (mm) (no pain) to 100 mm (worst pain imaginable). An increase in score indicates worsening pain, while a decrease represents a response to the intervention.
Change in VAS Stiffness Score from Baseline to Six Weeks | 6 weeks
  Stiffness scale ranges from 0 millimeters (mm) (no stiffness) to 100 mm (worst stiffness imaginable). An increase in score indicates worsening stiffness, while a decrease represents a response to the intervention.
Change in VAS Fatigue Score from Baseline to Six Weeks | 6 weeks
  Fatigue scale ranges from 0 millimeters (mm) (no fatigue) to 100 mm (worst fatigue imaginable)An increase in score indicates worsening fatigue, while a decrease represents a response to the intervention.
Change in FACIT-Fatigue Score from Baseline to Six Weeks | 6 weeks
  This 13-item scale assesses levels of fatigue during daily activities over the past seven days. Higher scores indicate less fatigue (score range = 0 - 52). Positive change scores indicate improved fatigue.

SECONDARY OUTCOMES:
Participant Satisfaction with Walk With Ease | 6 weeks
  This survey was designed by the Arthritis Foundation to assess participant satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Sheikh, MD, Principal Investigator — University of North Carolina, Chapel Hill; Leigh Callahan, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Katherine Kaufman, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Rheumatology Clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helmick CG, Felson DT, Lawrence RC, Gabriel S, Hirsch R, Kwoh CK, Liang MH, Kremers HM, Mayes MD, Merkel PA, Pillemer SR, Reveille JD, Stone JH; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part I. Arthritis Rheum. 2008 Jan;58(1):15-25. doi: 10.1002/art.23177. PMID 18163481
- [Background] Ward MM. Prevalence of physician-diagnosed systemic lupus erythematosus in the United States: results from the third national health and nutrition examination survey. J Womens Health (Larchmt). 2004 Jul-Aug;13(6):713-8. doi: 10.1089/jwh.2004.13.713. PMID 15333286
- [Background] Bartels CM, Buhr KA, Goldberg JW, Bell CL, Visekruna M, Nekkanti S, Greenlee RT. Mortality and cardiovascular burden of systemic lupus erythematosus in a US population-based cohort. J Rheumatol. 2014 Apr;41(4):680-7. doi: 10.3899/jrheum.130874. Epub 2014 Feb 15. PMID 24532834
- [Background] Bernatsky S, Boivin JF, Joseph L, Manzi S, Ginzler E, Gladman DD, Urowitz M, Fortin PR, Petri M, Barr S, Gordon C, Bae SC, Isenberg D, Zoma A, Aranow C, Dooley MA, Nived O, Sturfelt G, Steinsson K, Alarcon G, Senecal JL, Zummer M, Hanly J, Ensworth S, Pope J, Edworthy S, Rahman A, Sibley J, El-Gabalawy H, McCarthy T, St Pierre Y, Clarke A, Ramsey-Goldman R. Mortality in systemic lupus erythematosus. Arthritis Rheum. 2006 Aug;54(8):2550-7. doi: 10.1002/art.21955. PMID 16868977
- [Background] Lerang K, Gilboe IM, Steinar Thelle D, Gran JT. Mortality and years of potential life loss in systemic lupus erythematosus: a population-based cohort study. Lupus. 2014 Dec;23(14):1546-52. doi: 10.1177/0961203314551083. Epub 2014 Sep 10. PMID 25209070
- [Background] Trager J, Ward MM. Mortality and causes of death in systemic lupus erythematosus. Curr Opin Rheumatol. 2001 Sep;13(5):345-51. doi: 10.1097/00002281-200109000-00002. PMID 11604587
- [Background] Robb-Nicholson LC, Daltroy L, Eaton H, Gall V, Wright E, Hartley LH, Schur PH, Liang MH. Effects of aerobic conditioning in lupus fatigue: a pilot study. Br J Rheumatol. 1989 Dec;28(6):500-5. doi: 10.1093/rheumatology/28.6.500. PMID 2590802
- [Background] Daltroy LH, Robb-Nicholson C, Iversen MD, Wright EA, Liang MH. Effectiveness of minimally supervised home aerobic training in patients with systemic rheumatic disease. Br J Rheumatol. 1995 Nov;34(11):1064-9. doi: 10.1093/rheumatology/34.11.1064. PMID 8542209
- [Background] Ramsey-Goldman R, Schilling EM, Dunlop D, Langman C, Greenland P, Thomas RJ, Chang RW. A pilot study on the effects of exercise in patients with systemic lupus erythematosus. Arthritis Care Res. 2000 Oct;13(5):262-9. doi: 10.1002/1529-0131(200010)13:53.0.co;2-8. PMID 14635294
- [Background] Tench CM, McCarthy J, McCurdie I, White PD, D'Cruz DP. Fatigue in systemic lupus erythematosus: a randomized controlled trial of exercise. Rheumatology (Oxford). 2003 Sep;42(9):1050-4. doi: 10.1093/rheumatology/keg289. Epub 2003 Apr 16. PMID 12730519
- [Background] Clarke-Jenssen AC, Fredriksen PM, Lilleby V, Mengshoel AM. Effects of supervised aerobic exercise in patients with systemic lupus erythematosus: a pilot study. Arthritis Rheum. 2005 Apr 15;53(2):308-12. doi: 10.1002/art.21082. No abstract available. PMID 15818657
- [Background] Carvalho MR, Sato EI, Tebexreni AS, Heidecher RT, Schenkman S, Neto TL. Effects of supervised cardiovascular training program on exercise tolerance, aerobic capacity, and quality of life in patients with systemic lupus erythematosus. Arthritis Rheum. 2005 Dec 15;53(6):838-44. doi: 10.1002/art.21605. PMID 16342102
- [Background] Yuen HK, Holthaus K, Kamen DL, Sword DO, Breland HL. Using Wii Fit to reduce fatigue among African American women with systemic lupus erythematosus: a pilot study. Lupus. 2011 Oct;20(12):1293-9. doi: 10.1177/0961203311412098. Epub 2011 Jun 23. PMID 21700656
- [Background] Eriksson K, Svenungsson E, Karreskog H, Gunnarsson I, Gustafsson J, Moller S, Pettersson S, Bostrom C. Physical activity in patients with systemic lupus erythematosus and matched controls. Scand J Rheumatol. 2012 Aug;41(4):290-7. doi: 10.3109/03009742.2011.624117. Epub 2012 May 31. PMID 22651371
- [Background] Mancuso CA, Perna M, Sargent AB, Salmon JE. Perceptions and measurements of physical activity in patients with systemic lupus erythematosus. Lupus. 2011 Mar;20(3):231-42. doi: 10.1177/0961203310383737. Epub 2010 Dec 23. PMID 21183562
- [Background] Callahan LF, Shreffler JH, Altpeter M, Schoster B, Hootman J, Houenou LO, Martin KR, Schwartz TA. Evaluation of group and self-directed formats of the Arthritis Foundation's Walk With Ease Program. Arthritis Care Res (Hoboken). 2011 Aug;63(8):1098-107. doi: 10.1002/acr.20490. PMID 21560255